CLINICAL TRIAL: NCT05519618
Title: Multi-modality Evaluation of Flow Rate, Pressure and Size of Spine Epidural Venous Plexus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202112207RINC
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms; Spine Tumor; Venous Hypertension
Keywords: Spine tumor; Venous pressure; Internal vertebral venous plexus; Epidural venous plexus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patient planned to receive debulking or en bloc resection of vertebral tumor.
  Interventions: Procedure: Epidural veins pressure and flow measurement

INTERVENTIONS:
Procedure: Epidural veins pressure and flow measurement — The purpose of this study is to measure to pressure and flow of epidural venous plexus.
  The procedure will be performed alongside during pre-operative embolization at the angiography suite.
  It will be performed under general anesthesia. A the start of the procedure, a venous access will be established at the inguinal region. Co-axial catheters will be navigated to epidural venous plexus under the guidance of fluoroscopy. After the placement of catheter, the pressure and flow of epidural venous plexus will be measured at three time points: 1. Right after catheter reach the targeted location 2. Right before embolization. 3. After embolization. The participant will be instructed to control their breathe during measurement.
  After measurement, the catheter will be removed alongside with embolization devices, and achieved hemostasis as routine.

SUMMARY:
Vertebra is one of the most common site of metastatic disease, which may cause severe pain or neurological deficit. Debulking surgery usually has better local control and survival benefit as compared with decompression or radiotherapy. However, debulking surgery often accompany with massive blood loss, which may cause hemorrhagic shock or death. The major bleeding point during operation including tumor parenchyma, arteries that are difficult to ligate, and epidural venous plexus. Vascularity of tumor parenchyma had been associated with increased intraoperative blood loss, on the other hand, there is a lack in the literature regarding to evaluation of the size, flow and pressure of epidural venous plexus, and their changes after embolization.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who receive pre-operative angiography and possible embolization before debulking surgery or en bloc resection of the spinal tumor.
2. The tumor has to be located in thoracic or lumbar spine.

Exclusion Criteria:

1. Confirmed non-tumor diagnosis.
2. Patient who cannot tolerate the procedure due to severe pain.
3. Patients who cannot receive angiography or embolization due to contraindications, including poor renal function (Serum creatinine >2.0 deciliter/mg or estimated glomerular filtration rate(eGFR)) < 30ml/min) , severe allergy to contrast medium, uncorrectable coagulopathy and bleeding diathesis.
4. Patient who has severe neurological deficit that should receive emergent decompression.
5. Poor image quality.
6. Expected life expectancy < 6 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are suspected to have spine tumor, and referred to the multi-discipline spine oncology team in the study institute, for evaluation of debulking surgery or en bloc resection of the spinal tumor.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Epidural venous pressure | During the embolization intervention.
  Epidural venous pressure measured with pressure wire after reach the targeted location, before embolization and after embolization during the embolization procedure.
Epidural venous flow rate. | During the embolization intervention.
  Epidural venous flow rate measured with fluoroscopy after reach the targeted location, before embolization and after embolization during the embolization procedure.

SECONDARY OUTCOMES:
Size of epidural venous plexus. | During the embolization intervention.
  Measuring the size of epidural venous plexus with fluoroscopy after reach the targeted location, before embolization and after embolization during the embolization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: YuCheng Huang, M.D., Principal Investigator — Department of Radiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan